CLINICAL TRIAL: NCT06922331
Title: Age-Stratified Efficacy of Upadacitinib in Refractory Inflammatory Bowel Disease Among Asian Populations: Pediatric Crohn's Disease Versus Elderly Ulcerative Colitis Cohort Analysis
Brief Title: Upadacitinib for Refractory IBD in Asian Children and Elderly: Age-Stratified Analysis
Acronym: UPA-AGE
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jiayin Yao, Associate Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2025ZSLYEC-149
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Crohn's Disease (CD); Ulcerative Colitis (UC); Refractory Crohn's Disease; Refractory Ulcerative Colitis; Inflammatory Bowel Disease (IBD); Pediatric Crohn's Disease; Geriatric Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pediatric Crohn's Disease (CD) Group: Patients aged 9-17 years diagnosed with refractory Crohn's disease who received upadacitinib treatment.
  Interventions: Drug: Upadacitinib
- Elderly Ulcerative Colitis (UC) Group: Patients aged 60 years or older diagnosed with refractory ulcerative colitis who received upadacitinib treatment.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — A selective Janus kinase (JAK) 1 inhibitor used for the treatment of refractory inflammatory bowel disease.

SUMMARY:
This single-center, retrospective study aims to evaluate the effectiveness and safety of upadacitinib (UPA) in Asian pediatric patients with refractory Crohn's disease (CD) and elderly patients with refractory ulcerative colitis (UC). The study will analyze data from 21 patients (11 children aged 9-17 with CD and 10 adults aged 60 and older with UC) treated at the Sixth Affiliated Hospital of Sun Yat-sen University between January 2023 and December 2024. The primary objective is to assess the clinical remission rate and endoscopic response rate in both groups. Secondary objectives include comparing treatment outcomes between the two age groups, exploring the impact of immunosenescence on UPA efficacy in elderly UC patients, and analyzing the correlation between laboratory markers (CRP, albumin) and clinical outcomes. This study is the first in Asia to investigate the age-stratified efficacy of upadacitinib in pediatric CD and elderly UC patients. The findings will provide crucial real-world evidence to inform individualized treatment strategies for these specific populations. Patients included in this study will have previously failed at least two biological therapies. Data collected will include demographics, disease characteristics, prior treatment history, UPA dosage and duration, clinical and endoscopic scores (PCDAI/Mayo, SES-CD/UCEIS), imaging results, laboratory values, and adverse events. The study is registered on ClinicalTrials.gov (NCT06274996). Ethical considerations will be addressed through data anonymization and a waiver of informed consent due to the retrospective nature of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD according to the "Consensus on Diagnosis and Treatment of Inflammatory Bowel Disease (2023)"; Failure of at least two prior biological therapies (anti-TNF/anti-integrin/IL-12/23 inhibitors); Complete baseline and follow-up data (at least 12 weeks))

Exclusion Criteria:

* Active infection, malignancy, severe cardiovascular disease, or hepatic/renal insufficiency; Pregnancy or breastfeeding; Use of other JAK inhibitors within 30 days prior to baseline)

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Asian pediatric patients (ages 9-17) with refractory Crohn's disease and elderly patients (60 years and older) with refractory ulcerative colitis.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical Remission Rate at Week 12 | Week 12
  he proportion of patients achieving clinical remission at 12 weeks, as defined by [Specify the definition of clinical remission, e.g., "a Mayo score ≤ 2 with no individual subscore > 1" for UC or "a PCDAI score < 10" for CD].
Endoscopic Response Rate at Week 12 | Week 12
  The proportion of patients achieving endoscopic response at 12 weeks, as defined by [Specify the definition of endoscopic response, e.g., "a decrease of ≥50% from baseline in the SES-CD score" for CD or "a decrease of ≥ 1 point from baseline in the UCEIS" for UC].

SECONDARY OUTCOMES:
Clinical Response Rate at Week 12 | Week 12
  The proportion of patients achieving clinical response at 12 weeks, as defined by [Specify the definition of clinical response, e.g., "a decrease of ≥ 3 points from baseline in the Mayo score" for UC or "a decrease of ≥ 20 points from baseline in the PCDAI score" for CD].
Change in CRP from Baseline to Week 12 | Baseline to Week 12
  The change in C-reactive protein (CRP) levels from baseline to 12 weeks after treatment initiation.

OTHER OUTCOMES:
Incidence of Adverse Events | Week 0 to Week 12
  The number and type of adverse events occurring during the 12-week treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No